CLINICAL TRIAL: NCT01997853
Title: Effect of Scaling & Root Planing (SRP) Combined With Therapy Of Omega-3 Fatty Acid on Clinical Parameters and Serum Levels of C-Reactive Protein (CRP) in Chronic Periodontitis - A Randomised Control Trial.
Brief Title: Omega-3 Fatty Acids in Chronic Periodontitis.
Acronym: omega3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, GIRISH DEORE, Principal Investigator, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TKDC13
Record Dates: First submitted 2013-11-20; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Periodontitis
Keywords: Omega 3 fatty acids; C Reactive Protein; Host Modulation; Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Group (Active Comparator): Patients with Chronic Periodontitis in Test Group were prescribed Omega 3 fatty acid tablets 300mg once daily for 12 weeks
  Interventions: Drug: Omega 3 fatty acid
- Control Group (Placebo Comparator): Patients with Chronic Periodontitis in Control Group were prescribed Placebo tablets once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega 3 fatty acid — Patients with Chronic Periodontitis in Test Group were prescribed Omega 3 fatty acid tablets 300mg once daily for 12 weeks and SRP at baseline
  Other Names: Mega-3
  Arms: Test Group
Drug: Placebo — Patients with Chronic Periodontitis in Control Group were prescribed Placebo tablets once daily for 12 weeks and SRP
  Arms: Control Group

SUMMARY:
Omega 3 fatty acids is one such dietary supplement, known to modulate the host response in chronic conditions like cardiovascular diseases, rheumatoid arthritis, ischemic cerebrovascular diseases, osteoporosis by producing Resolvins and protectins without showing any inadvertent effects.Addition of systemic Omega 3 Fatty Acids with SRP may enhance the therapeutic result of Chronic Periodontitis owing to host modulation & anti-inflammatory properties. If proven, this can be used as a routine treatment modality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients within age group of 30 to 55 years.
2. Systemically healthy individuals.
3. Patients with chronic generalized periodontitis (moderate and severe)according to Center for Disease Control (CDC) working group, 2007 criteria.

Exclusion Criteria:

1. Patients with systemic illnesses (i.e., diabetes mellitus, cancer, human immunodeficiency syndrome, bone metabolic diseases, or disorders that compromise wound healing, radiation, or immunosuppressive therapy),
2. Smoking,
3. Chronic alcoholics,
4. Pregnancy or lactation,
5. Use of Non Steroidal Anti Inflammatory Drugs, steroids or antibiotics / antimicrobials within September 2012 to August 2013,
6. Confirmed or suspected intolerance to omega 3 fatty acids,
7. Periodontal therapy done within the September 2012 to August 2013.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum CRP level at 6 weeks and 12 weeks | baseline, 6 weeks, 12 weeks
  changes from baseline in biochemical parameter, serum CRP levels were assessed at 6 weeks and 12 weeks after starting therapy with omega 3 fatty acids. Serum CRP level was measured in milligram/liter (mg/l)
Changes from baseline in pocket depth (PD) at 6 weeks and 12 weeks | baseline, 6 weeks and 12 weeks
  changes from baseline in clinical parameter, PD were assessed at 6 weeks and 12 weeks after starting therapy with omega 3 fatty acids. PD was measured in millimeter.
Changes from baseline in Clinical Attachment Level (CAL) at 6 weeks and 12 weeks. | baseline, 6 weeks and 12 weeks
  changes from baseline in clinical parameter, CAL were assessed at 6 weeks and 12 weeks after starting therapy with omega 3 fatty acids. CAL was measured in millimeter.

SECONDARY OUTCOMES:
Changes from baseline in Gingival Index (GI) at 6 weeks and 12 weeks | baseline, 6 weeks and 12 weeks
  changes from baseline in standard clinical parameter, GI were assessed at 6 weeks and 12 weeks after starting therapy with omega 3 fatty acids. GI has a scoring criteria specified by Silness & Loe, 1963.
Changes from baseline in Plaque Index (PI) at 6 weeks and 12 weeks | baseline, 6 weeks and 12 weeks
  changes from baseline in standard clinical parameter, PI were assessed at 6 weeks and 12 weeks after starting therapy with omega 3 fatty acids. PI has a scoring criteria specified by Loe & Silness, 1964.
Changes from baseline in Oral Hygiene Index Simplified (OHIS) at 6 weeks and 12 weeks. | baseline, 6 weeks and 12 weeks
  changes from baseline in standard clinical parameter, OHIS were assessed at 6 weeks and 12 weeks after starting therapy with omega 3 fatty acids. OHIS has a scoring criteria specified by Greene and Vermilion, 1964.
Changes from baseline in Sulcus Bleeding Index (SBI) at 6 weeks and 12 weeks | baseline, 6 weeks and 12 weeks
  changes from baseline in standard clinical parameter, SBI were assessed at 6 weeks and 12 weeks after starting therapy with omega 3 fatty acids. SBI has a scoring criteria specified by Muhleman (1971).

CONTACTS AND LOCATIONS:
Overall Officials: Girish D Deore, BDS, Principal Investigator — Post Graduate Student
Locations (1):
- Tatyasaheb Kore Dental College and Research Centre, New Pargaon, Kolhāpur, Maharashtra, India